CLINICAL TRIAL: NCT02419261
Title: Assessment of Sensory and Motor Blockade of the Adductor Canal Blockade Performed for Surgery of Arthroscopic Anterior Cruciate Ligament Repair
Brief Title: Assessment of Adductor Canal Blockade in Anterior Cruciate Ligament Surgery
Acronym: ACB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, J P Lecoq, MD, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gauthier - Lecoq - Goffin
Record Dates: First submitted 2015-04-02; First posted 2015-04-17 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Surgery of Arthroscopic Anterior Cruciate Ligament Repair
Keywords: knee surgery; anterior cruciate ligament surgery; nerve block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adductor Canal Blockade (Active Comparator): In this group, patient will benefit of an ultrasound guided adductor canal blockade (20 ml of Ropivacaine 0.75%) as analgesic nerve blockade for their surgery of anterior cruciate ligament repair
  Interventions: Drug: Analgesic nerve blockade (Ropivacaine); Procedure: Arthroscopic surgical repair of the anterior cruciate ligament
- Femoral Nerve Blockade (Active Comparator): In this group, patient will benefit of an ultrasound guided femoral nerve blockade (20 ml of Ropivacaine 0.75%) as analgesic nerve blockade for their surgery of anterior cruciate ligament repair
  Interventions: Drug: Analgesic nerve blockade (Ropivacaine); Procedure: Arthroscopic surgical repair of the anterior cruciate ligament

INTERVENTIONS:
Drug: Analgesic nerve blockade (Ropivacaine) — Analgesic nerve blockade for Arthroscopic surgical repair of the anterior cruciate ligament
Procedure: Arthroscopic surgical repair of the anterior cruciate ligament

SUMMARY:
Assessment of sensory and motor blockade of adductor canal blockade performed for anterior cruciate ligament repair in comparison with femoral nerve blockade.

DETAILED DESCRIPTION:
The adductor canal blockade is a reliable technique for analgesia after knee surgery. It is a safe technique, avoiding muscle weakness, and by this way limiting the risk of fall. Injection of local anaesthetics in the adductor canal does not block the sole saphenous nerve. Demonstration of a proximal spreading, around the branches of the femoral nerve have been made. The aim of this study is to assess a possible spreading from the adductor to the the popliteal fossa, where sciatic nerve and its branches are located. Pinprick test all around the knee and the leg, combined with motor assessment of the muscle of the leg and the ankle will be realised. This assessment was compared with femoral nerve blockade, classically used for analgesia after this kind of surgery (anterior cruciate ligament repair)

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for anterior cruciate ligament repair

Exclusion Criteria:

* Refusal to study,
* coagulation disorder,
* infection at the puncture site,
* preexisting neuropathy,
* allergy to local anesthetics,
* renal or hepatocellular insufficiency,
* context of chronic pain,
* drugs abuse,
* pregnant patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Cold sensitivity assessment (cold, very cold, no sensation) | From 30 to 60 minutes after nerve blockade
  sensitivity description (cold, very cold, no sensation)
Motor blockade assessment (dynamometer) | From 30 to 60 minutes after nerve blockade
  motor blockade evaluation with dynamometer

SECONDARY OUTCOMES:
Postoperative pain assessment (visual analgesic scale) | At 2, 4, 6 postoperative hours
  Evaluation with visual analgesic scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre H Lecoq, MD PhD, Principal Investigator — University of Liege, University Hospital
Locations (1):
- University of Liege, University Hospital, Liège, Belgium